CLINICAL TRIAL: NCT01794078
Title: A Randomized, 4-Sequence, Double-Blind Study to Test the Safety of Combined Dosing With Aminophylline and Ambrisentan in Exercising Healthy Human Volunteers at Simulated High Altitude
Brief Title: A Study to Test the Safety of Combined Dosing With Aminophylline and Ambrisentan in Exercising Healthy Human Volunteers at Simulated High Altitude
Acronym: GQ02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert J Noveck, M.D. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Robert J Noveck, M.D., Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00037605
Record Dates: First submitted 2013-02-10; First posted 2013-02-18 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Acute Mountain Sickness and Fatigue
Keywords: Acute Mountain Sickness; High altitude induced fatigue
MeSH Terms: conditions — Altitude Sickness; Fatigue | interventions — Aminophylline; Ethylenediamines; ambrisentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- Control (Placebo Comparator): Oral placebo, administered as single dose during simulated altitude episodes Cycle 1 and Cycle 2
  Interventions: Other: Placebo
- Aminophylline 400 mg (Experimental): Oral aminophylline 400 mg, administered as single dose during simulated altitude episodes Cycle 1 and Cycle 2
  Interventions: Drug: Aminophylline 400 mg
- ambrisentan 5 mg (Experimental): Oral ambrisentan 5 mg, administered as single dose during simulated altitude episodes Cycle 1 and Cycle 2
  Interventions: Drug: Ambrisentan 5 mg
- Combined aminophylline 400 mg and ambrisentan 5 mg (Experimental): Oral combined aminophylline 400 mg and ambrisentan 5 mg, administered as single doses during simulated altitude episodes Cycle 1 and Cycle 2
  Interventions: Drug: Aminophylline 400 mg; Drug: Ambrisentan 5 mg

INTERVENTIONS:
Drug: Aminophylline 400 mg — Xanthine derivative
  Other Names: Mixture of theophylline and ethylene diamine
  Arms: Aminophylline 400 mg; Combined aminophylline 400 mg and ambrisentan 5 mg
Drug: Ambrisentan 5 mg — Endothelin receptor antagonist
  Other Names: Letairis; Volibris
  Arms: Combined aminophylline 400 mg and ambrisentan 5 mg; ambrisentan 5 mg
Other: Placebo
  Arms: Control

SUMMARY:
Acute exposure of the unacclimatized human body to high altitude leads to health complications, such as loss of exercise performance capacity and fatigue. The investigators have found that the combination of the xanthine drug theophylline and the endothelin receptor antagonist ambrisentan improves the exercise performance capacity of rats under simulated high altitude. In young, healthy human volunteers, this combination of drugs has not increase toxicity over the single compounds under sea-level conditions. The aim of this study is to test whether the combination of theophylline, supplied as its more soluble formulation aminophylline, and ambrisentan, are also safe to take under simulated high altitude of 4,267 meters, under both resting and exercising conditions. The study also aims to test whether this drug combination improves exercise capacity in humans. In this study, human subjects will be randomized to one of four treatment sequences and receive the same study drug(s) throughout all procedures. The study consists of an initial exercise test, followed by two cycles of drug testing at simulated high altitude: Cycle 1 - resting subjects receiving study drug at simulated altitude and continually monitored for safety with pharmacodynamic and pharmacokinetic assessments; and Cycle 2, the same as Cycle 1, with the addition of exercise testing. It is hypothesized that the combination of aminophylline and ambrisentan is not only safe under simulated high altitude, but also improves exercise performance capacity, in comparison with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give written Informed Consent to participate in the study prior to undergoing any screening procedures. The subject will be given a signed and dated copy of the Informed Consent.
* Subjects must be healthy non-smoking (for 6 months or greater at commencement of Cycle 1) adult male and female volunteers; at least 18 through 50 years at screening, with a BMI of 18-33 kg/m2 and weighing at least 143 lbs. (65 kg). Subjects' health status will be determined by the medical history, physical examination, vital signs, ECG, blood chemistry, hematology, and urinalysis performed at screening.
* Subjects must be willing to fast a minimum of 2 hours prior to screening.
* Subjects must be willing to abstain from alcohol and xanthine-containing food and beverages from 48 hours before check-in for each study day,
* Women who are of non-childbearing potential, must be:
* Surgically sterile (removal of both ovaries and/ or uterus at least 12 months prior to dosing) and with an FSH level at screening of ≥ 40 mIU/mL.
* Naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to dosing on Day -1, and with an FSH level at screening of ≥ 40 mIU/mL.
* Women of child-bearing potential must have a negative serum or urine pregnancy test at screening, during the study, and must agree to avoid pregnancy during study and for three months after the last dose of study drug. Pregnancy is tested at screening, during check-in of each testing cycle, during the follow-up visit, and at any given point if deemed necessary to the PI or designate. During treatment, women of child-bearing potential must use two acceptable methods of contraception at the same time unless the subject has had a documented tubal sterilization or chooses to use a Copper T 380A IUD or LNG 20 IUS, in which case no additional contraception is required. Abstinence is not considered a form of contraception. Medically acceptable contraceptives include: (1) documented surgical sterilization (such as a hysterectomy), (2) barrier methods (such as a condom or diaphragm) used with a spermicide, or (3) an intrauterine device (IUD) or intrauterine system (IUS).
* Male subjects must agree to take all necessary measures to avoid causing pregnancy in their sexual partners during the study and for three months after the last dose of study drug. Medically acceptable contraceptives include: (1) surgical sterilization (such as a vasectomy), or (2) a condom used with a spermicidal. Contraceptive measures such as Plan B (TM), sold for emergency use after unprotected sex, are not acceptable methods for routine use.
* Subjects must agree not to donate blood, platelets, or any other blood components 30 days, or plasma 90 days, prior to consenting and for 1 month after the last dose.
* Male subjects must agree not to donate sperm during the study and for 12 weeks after the last dose.

Exclusion Criteria:

* Subjects with laboratory results outside the normal range, if considered clinically significant (CS) by the PI or delegate. In addition, subjects must have a hemoglobin concentration of ≥ 12.0 g/dL.
* A mental capacity that is limited to the extent that the subject cannot provide legal consent or understand information regarding the side effects of the study drug.
* Currently abusing drugs or alcohol or with a history of drug or alcohol abuse within the past two years.
* Unwillingness or lack of ability to comply with the protocol, or to cooperate fully with the PI and site personnel.
* Use of any of the following:
* Any concomitant medication including oral contraceptive hormones. Subjects who have received any prescribed or non-prescribed (over-the-counter [OTC]) systemic medication, topical medications, or herbal supplements within 14 days from Day 1. St. John's Wort (hypericin) must not have been taken for at least 30 days prior to Cycle 1, Day 1.
* Any drugs, foods or substances known to be strong inhibitors or strong inducers of CYP enzymes (also known as cytochrome P450 enzymes); especially CYP 1A2, or Pgp within 7 days prior to Cycle 1, Day 1.
* Clinically significant ECG abnormality in the opinion of the PI or delegate.
* Vital signs or clinically significant laboratory values at the screening visit that in the opinion of the PI or delegate would make the subject an inappropriate candidate for the study.
* A VO2 max value of less than 42 mL/kg/min, as determined during exercise testing at screening. This value represents an educated estimate, and may be changed, to include new information, at the discretion of the PI.
* A history of, or otherwise indicated predisposition for, claustrophobia, i.e. the fear of closed, narrow spaces (because of the limited size of the high altitude chamber).
* A history of "undeserved" altitude sickness, i.e. altitude sickness at only moderate altitude. This would consist of altitude-related headaches, dizziness, or nausea during plane rides, or when traveling to moderately elevated locations of less than 2,743.2 meters/ 9,000 ft
* Has taken any other investigational drug during the 30 days prior to the screening visit or is currently participating in another investigational drug clinical trial.
* Made any significant donation or have had a significant loss of blood within 30, or donated plasma within 90 days of consenting.
* Receipt of a transfusion or any blood products within 90 days prior to commencement of Cycle 1
* History or manifestation of clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematologic or other medical disorders. For the purpose of the study, individual fitness and health are more important than family history of disease burden as a criterion for participation. For example, an individual may have significant family history of cardiovascular disease; however, the individual subject's active lifestyle makes a manifestation of such disease at young ages unlikely. To account for such expected variation, the ultimate decision whether to exclude or include an individual based on family history or manifestation of disease will be made by the PI. The PI may choose to use physiological assessments, such as e.g. ECG, blood pressure, and VO2 max fitness level as an aid for decision making.
* Any condition that might interfere with the absorption of the study medications or influence the interpretation of the results of the study.
* Subjects who are carriers of the Hepatitis B surface antigen (HbsAg), Hepatitis C antibody, or HIV antibody.
* Serious mental or physical illness within the past year.
* Male subjects who consume more than 28 units of alcohol per week and female subjects who consume more than 21 units of alcohol per week (one unit of alcohol equals 250 mL of beer, 100 mL of a medium glass of wine, or 25 mL of spirits) or those subjects who have a significant history of alcoholism or drug/ chemical abuse within the last 2 years.
* Failure to agree to abstain from alcohol, cola, tea, coffee, chocolate and other caffeinated drink/ food from 48 h before check-in for Cycles 1 & 2.
* Subjects who have used tobacco products or nicotine-containing products (including smoking cessation aids, such as gums or patches) within 6 months prior to commencement of Cycle 1
* Women of childbearing potential who are pregnant (as based on test results) or are breast feeding
* Subjects who have a history of hypersensitivity or idiosyncratic reaction to any of the products administered during the study.
* Subjects who, in the opinion of the PI (or delegate), should not participate in the study.
* Subjects who are employed by the Duke Clinical Research Unit and/or the Duke Hypobaric/ Hyperbaric Center
* Subjects who have a history of unexplained syncope or fainting from the collection of blood; i.e., autonomic dysfunction.
* Subjects who have a history of hypotension, including orthostatic hypotension. The ultimate decision about exclusion or inclusion of a potential subject is made by the PI.
* Lack of ability to understand verbal and/ or written English.
* History of clinically significant illness within 4 weeks prior to commencement of Cycle 1. In case a subject develops an illness between any of the study activities (Screening, Cycle 1, and Cycle 2), the subject may be removed from the study, if it deems appropriate and/ or necessary to the PI.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The safety of combined or single-dose aminophylline and ambrisentan at simulated high altitude in resting human subjects | Safety endpoints will be measured during an episode of simulated high altitude (Cycle 1), at least 7 days post screening
  Incidence and severity of Adverse Events, blood pressure, heart rate, ECGs, blood oxygen saturation (pulse oximetry), symptoms related to early acute mountain sickness (AMS)
The safety of combined or single-dose aminophylline and ambrisentan at simulated altitude in exercising human subjects | Safety endpoints will be measured during simulated high altitude (Cycle 2) at least 22 days post screening
  Incidence and severity of Adverse Events, blood pressure, heart rate, ECGs, blood oxygen saturation (pulse oximetry), symptoms related to acute mountain sickness (AMS)

SECONDARY OUTCOMES:
The efficacy of combined aminophylline and ambrisentan to improve exercise capacity under simulated high altitude | Drug effects on exercise capacity are assessed during an episode of simulated high altitude (Cycle 2), at least 22 days after screening
  Exercise capacity is measured as the self-chosen level of exercise burden during cycling on a bicycle ergometer
The influence of simulated high altitude on pharmacokinetic profiles and drug interaction of aminophylline and ambrisentan | Blood samples for drug interaction analysis are acquired during an episode of simulated high altitude (Cycle 1), at least 7 days past screening
  PK profiles will be compared between combined and single-dosed subjects

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Noveck, MD, PhD, Principal Investigator — Duke University; Claude A Piantadosi, MD, Study Director — Duke University; Thies Schroeder, PhD, Study Director — Duke University
Locations (2):
- United States (2):
  - Duke Center for Hyperbaric Medicine, Durham, North Carolina
  - Duke Clinical Research Unit (DCRU), Durham, North Carolina